CLINICAL TRIAL: NCT00774657
Title: Patterns Of Left Ventricular Remodeling In Patients With Aortic Stenosis Assessed By Two-Dimensional And Three-Dimensional Echocardiography
Brief Title: Ventricular Remodeling In Patients With Aortic Stenosis Assessed Echocardiography
Status: Withdrawn | Type: Observational
Why Stopped: Unable to identify and recruit suitable study subjects
Sponsor: Lahey Clinic (Other)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-090
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis; Valvular heart disease; Heart disease; Cardiovascular disease; Two dimensional echocardiography; Three dimensional echocardiography
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This preliminary study will compare the effectiveness of two-dimensional and three-dimensional echocardiographic measurements of wall thickness and left ventricular mass in patients with Aortic Stenosis

DETAILED DESCRIPTION:
This study will evaluate left ventricular patterns of remodeling and hypertrophy in patients with aortic stenosis, and compare two-dimensional echocardiography measurements (wall thickness) with three-dimensional echocardiography data(left ventricular mass). Along with a second objective to assess Doppler diastolic filling indices associated with the various patterns of left ventricular remodeling.

Previous studies(see reference list) were primarily derived from two-dimensional echo data set(based on wall thickness). Various patterns of left ventricular remodeling have been described in response to increased pressure overload.

Three-dimensional echocardiography is a relatively new technique that is being increasingly used in the Echocardiography Lab in selected patients. This technique holds promise of being more accurate for volume-related measurements than the standard 2-dimensional echocardiography techniques.

ELIGIBILITY:
Inclusion Criteria:

* Subjects more than 18 yrs of age through 90 yrs of age
* Both male and female
* Patients with moderate or severe isolated Aortic Stenosis
* Patients who have been referred for both two-dimensional and three- dimensional echocardiographies.

Exclusion Criteria:

* Poor acoustic windows
* h/o CAD and wall motion abnormality

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lahey Clinic patients who have been referred to the echocardiography lab for clinical indications, found to have a aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evaluate 2-dimensional and 3-dimensional echocardiography for LV patterns of remodeling and hypertrophy | 1 hour

SECONDARY OUTCOMES:
Assess doppler diastolic filling indices for patterns of LV remodeling | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sherif B. Labib, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Faggiano P, Rusconi C, Ghizzoni G, Sabatini T. Left ventricular remodeling and function in adult aortic stenosis. Angiology. 1994 Dec;45(12):1033-8. doi: 10.1177/000331979404501206. PMID 7985830
- [Background] Kupari M, Turto H, Lommi J. Left ventricular hypertrophy in aortic valve stenosis: preventive or promotive of systolic dysfunction and heart failure? Eur Heart J. 2005 Sep;26(17):1790-6. doi: 10.1093/eurheartj/ehi290. Epub 2005 Apr 28. PMID 15860517
- [Background] Salcedo EE, Korzick DH, Currie PJ, Stewart WJ, Lever HM, Goormastic M. Determinants of left ventricular hypertrophy in patients with aortic stenosis. Cleve Clin J Med. 1989 Sep;56(6):590-6. doi: 10.3949/ccjm.56.6.590. PMID 2530009
- [Background] Jenkins C, Bricknell K, Hanekom L, Marwick TH. Reproducibility and accuracy of echocardiographic measurements of left ventricular parameters using real-time three-dimensional echocardiography. J Am Coll Cardiol. 2004 Aug 18;44(4):878-86. doi: 10.1016/j.jacc.2004.05.050. PMID 15312875